CLINICAL TRIAL: NCT04607642
Title: A Randomized, Blinded, Placebo Controlled Phase 2 Trial of Concurrent Radiation Therapy and Cisplatin With and Without BMX-001 in Patients With Locally Advanced Head and Neck Cancer
Brief Title: Trial of BMX-001 or Placebo in Head and Neck Cancer Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Will be conducted as a different study with different sponsorship
Sponsor: BioMimetix JV, LLC (Industry)
Collaborators: Duke University (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMX-HN-201
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Head and Neck Cancer
Keywords: head and neck squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Mn(III) meso-tetrakis(N-n-butoxyethylpyridinium-2-yl)porphyrin; Radiotherapy; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded as well as use of blinded assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A BMX-001 (Experimental): Patients will receive standard of care radiation therapy plus Cisplatin. BMX-001 will be given by subcutaneous injection with a loading dose of 28 mg/subject given within 4 days prior to initiation of radiation therapy and followed by biweekly maintenance doses at half the loading dose for a total of 8 weeks.
  Interventions: Drug: BMX-001; Radiation: Radiation Therapy; Drug: Cisplatin
- B Placebo (Placebo Comparator): Patients will receive standard of care radiation therapy plus Cisplatin. Placebo will be given by subcutaneous injection with a loading dose of 28 mg/subject given within 4 days prior to initiation of radiation therapy and followed by biweekly maintenance doses at half the loading dose for a total of 8 weeks.
  Interventions: Radiation: Radiation Therapy; Drug: Cisplatin; Other: Placebo

INTERVENTIONS:
Drug: BMX-001 — BMX-001 consists of a porphyrin ring with pyridyl groups attached at each of the four methane bridge carbons. The nitrogen in the pyridyl ring is at the 2 position and has a side chain consisting of six carbons with an ether linkage. A manganese atom is chelated into the porphyrin ring and is the active center of the molecule. This molecule is an enzymatic scavenger of free radical species operating at close to diffusion-limited rates.
  Other Names: manganese butoxyethyl pyridyl porphyrin; MnTnBuOE-2-PyP5+
  Arms: A BMX-001
Radiation: Radiation Therapy — Treatment plan should include a continuous course of treatment delivered as single daily fractions of 2.0 to 2.1 Gy with a cumulative radiation dose between 60 Gy and 70 Gy. Planned radiation treatment volumes must include at least two oral mucosal sub-sites (buccal mucosa, retromolar trigone, floor of mouth, tongue, soft palate, hard palate) with a portion of each site receiving at least 50 Gy.
Drug: Cisplatin — Cisplatin is an IV chemotherapeutic agent approved to treat head and neck cancers. Cisplatin will be administered per institution's standard of care practice. Common standard of care practice includes dosing cisplatin at 100mg/m2 IV q21 days starting on Day 1 of RT for 2-3 doses or dosing cisplatin at 40 mg/m2 IV each week of RT for 6-7 total doses. Cisplatin will be infused per institutional guidelines.
Other: Placebo — The placebo to be used in this study is 0.9% Sodium Chloride Injection, USP.
  Arms: B Placebo

SUMMARY:
There are an estimated 65,000 newly diagnosed cases of head and neck cancer each year in the United States. The most common treatment for head and neck cancers is radiotherapy in combination with cisplatin chemotherapy. This treatment regimen is effective in killing the tumor; however, the normal tissues that line the mouth and throat can sustain severe injury from the radiation. Side-effects incurred during irradiation include: mucositis, xerostomia, swelling, trouble swallowing, pain, infections, cavities, hair loss and reddening of the skin. Some of these side effects can be so severe that patients require feeding tubes and management of severe pain can lead to the premature halt of radiotherapy. There are currently no effective radio-protectors used to ameliorate these severe side-effects.

BioMimetix has developed small molecular weight superoxide dismutase (SOD) mimetic, BMX-001, that is a very potent radio-protector of head and neck tissues. In our first clinical trial in a head and neck cancer patient cohort using this drug, we have early evidence that BMX-001 may protect against radiation-induced mucositis and xerostomia.

This will be a randomized, placebo-controlled Phase 2 clinical trial to study the effects of BMX-001 (14 mg/subject biw) + radiation therapy + cisplatin against placebo + radiation therapy + cisplatin in prevention of acute and chronic mucositis and xerostomia.

DETAILED DESCRIPTION:
This study will seek to confirm protection of normal tissues by assessing the incidence, severity and duration of mucositis in a randomized, placebo controlled, Phase 2 clinical trial of BMX-001 in combination with standard RT and chemotherapy in newly diagnosed head and neck cancer patients (162 subjects, 1:1 randomization study drug: placebo).

The study will also confirm protection of normal tissues by assessing the acute and chronic extent of xerostomia in the same trial.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed (histologically or cytologically) diagnosis of squamous cell carcinoma of the oropharynx, larynx, hypopharynx, nasopharyngeal, or oral cavity with clinical or pathologic high-risk features who will be receiving radiation and concurrent cisplatin chemotherapy.
2. Treatment plan to receive a continuous course of IMRT delivered as single daily fractions of 2.0 to 2.1 Gy with a cumulative radiation dose between 60 Gy and 70 Gy depending on whether patients are receiving post-operative or definitive intent therapy respectively.
3. For patients undergoing curative intent resection, Patients must have undergone gross total surgical resection within 56 days prior to registration and beginning of therapy under the clinical trial.
4. General history and physical examination by a qualified head and neck cancer specialist and physician within 8 weeks prior to enrollment (including fiberoptic endoscopy).
5. Axial imaging of the neck and chest- CT, MRI and/or PET/CT is acceptable, within 8 weeks prior to date of consent.
6. Age ≥ 18 years.
7. Zubrod Performance Status 0-2 within 4 weeks prior to enrollment.
8. CBC/differential obtained within 2 weeks prior to starting the study drug with adequate bone marrow function
9. Adequate hepatic function
10. Adequate renal function defined as follows:
11. Patient must be willing and able to follow study procedures and instructions.
12. Patient must provide study-specific informed consent within 28 days prior to starting the study drug.
13. Negative pregnancy test for women of child-bearing potential within 48 hours prior to first dose of BMX-001.
14. Women of childbearing potential and male participants must agree to use a medically effective means of birth control throughout their participation in the treatment phase of the study and until 12 months following the last study treatment.

Exclusion Criteria:

1. Distant metastasis
2. Hypertension
3. Grade ≥2 hypotension at screening
4. Concurrent treatment with nitrates or other drugs that may, in the judgment of the treating investigator, create a risk for a precipitous decrease in blood pressure
5. History of syncope within the last 6 months
6. Patients receiving, or unable to stop use of prohibited medications
7. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
8. Women who are breast feeding are not eligible
9. Known hypersensitivity to compounds of similar chemical composition to BMX-001
10. Grade 3-4 electrolyte abnormalities (CTCAE v 5.0)
11. Prior unrelated malignancy requiring current active treatment with exceptions
12. Prior history of HNSCC receiving radiation or chemo-radiation.
13. Prior systemic chemotherapy for the study cancer (including neoadjuvant chemotherapy); note that prior chemotherapy for a different cancer is allowable.
14. Prior radiotherapy that would result in overlap of radiation treatment fields with planned treatment for study cancer.
15. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >480 milliseconds (ms) using the specific/usual choice by clinical center for correction factor.
16. A history of additional risk factors for TdP
17. Severe, active co-morbidity as defined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Mucositis Incidence | 12 weeks
  The primary outcome measure used for each study subject is a dichotomous measure of whether they experienced severe oral mucositis (OM, defined as grade 3 or 4 according to WHO criteria) at any time between the first IMRT fraction until 30 days after the completion of RT. The primary analysis will thus test the difference in the proportion of subjects from each treatment group who experience severe OM.

SECONDARY OUTCOMES:
Mucositis Duration | 12 weeks
  The interval (measured in days) from the date of first determination of severe OM to the date of the first determination of not having severe OM, without a subsequent instance of severe OM.
Mucositis Severity | 12 weeks
  Days it takes for patients in each arm to develop severe oral mucositis.
Xerostomia Incidence | 1, 6, 12, and 24 months
  The dichotomous measure of whether the study subject had grade 2 (or greater) Xerostomia (as defined by CTCAE v 5.0). This will be assessed at 1, 6, 12, and 24 months after completion of RT.
Saliva Production Measurements | 1, 6, 12, and 24 months
  The continuous measure of saliva production (g/min), measured at baseline and 1, 6, 12, and 24 months after completion of RT. Both stimulated and unstimulated saliva production will be measured.
Radiation Dermatitis Duration | 12 weeks
  The continuous endpoint of duration of radiation dermatitis, where duration is defined as the interval (measured in days) from the date of first determination of radiation dermatitis to the date of the first determination of not having radiation dermatitis, without a subsequent instance of radiation dermatitis. For any subject whose radiation dermatitis persists, the final date will be 30 days after the completion of RT.
Overall Survival | 2 years
  Overall survival (OS), defined as the interval (measured in days) from the date of randomization until the date of death from any cause.
Disease Free Survival | 2 years
  Disease-free survival (DFS), defined as the interval (measured in days) from the date of randomization until the date of CT scan showing tumor progression.

CONTACTS AND LOCATIONS:
Overall Officials: James Crapo, MD, Study Director — BioMimetix JV, LLC

IPD SHARING:
Plan to Share IPD: No